CLINICAL TRIAL: NCT02848898
Title: The Effects of Focal Vibration on Central and Peripheral Spasticity in Multiple Sclerosis Patients. A Randomized, Multicenter, Double Blinded vs Placebo Study
Brief Title: The Effects of Focal Vibration on Spasticity in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Emanuele Spina, Resident, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 71/15
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis
Keywords: Focal Vibrations; Neurorehabilitation; Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Equistasi Group (Experimental): arm treated with application of devices
  Interventions: Device: Equistasi
- Placebo Group (Placebo Comparator): arm treated with application of inactivated devices
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Equistasi
  Arms: Equistasi Group
Other: Placebo
  Arms: Placebo Group

SUMMARY:
This trial consists of application of little devices (named Equistasi®) generating focal vibrations to treat spasticity in neurological patients, affected by multiple sclerosis. The expected effects are on gait and postural instability.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis affected
* Spasticity
* EDSS (Expanded Disability Status Scale) 0 - 5,5
* Patients able to sign informed consent

Exclusion Criteria:

* Age less than 18 years old and more than 65 years old
* Pacemaker
* Pregnancy
* Comorbidities as: cancer, hypertension not controlled by drugs
* concurrent therapies with antidepressant or corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Gait Velocity | one year
  evaluation of gait velocity in m/s
First step length | one year
  first step length in cm
Swing phase | one year
  swing phase measured in seconds
Stance phase | one year
  stance phase measured in seconds
Double support time | one year
  double support time measured in seconds

SECONDARY OUTCOMES:
H/M ratio | one year
  evaluation of neurophysiological modifications in treated patients vs placebo group, as ratio between H max and M max in tibial posterior nerve, in Unit
Berg Balance Scale | one year
  Evaluation of balance with a self administered scale, measured in Unit
Modified Fatigue Scale | one year
  evaluation of fatigue with a self administered scale, measured in Unit

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Giuseppe Orefice, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No